CLINICAL TRIAL: NCT06912074
Title: Comparing Hypofractionated Concurrent Chemoradiotherapy Versus Conventional Fractionated Concurrent Chemoradiotherapy Following Induction Chemo-immunotherapy in Patients With Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma: A Prospective, Open-Label, Randomized Phase II Clinical Trial
Brief Title: Hypofractionated vs. Conventional Chemoradiotherapy After Induction Chemo-immunotherapy for Unresectable Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10127
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Esophageal Squamous Cell Carcinoma; Hypofractionated Concurrent Chemoradiotherapy; Conventional Fractionated Concurrent Chemoradiotherapy; Induction chemoimmunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated CCRT group (Experimental): All patients will receive hypofractionated radiotherapy once daily, five days per week, followed by a boost. Three weeks after the completion of the first phase of hypofractionated radiotherapy, tumor response and cardiopulmonary function will be evaluated. For patients who achieve a partial response, have no deep esophageal ulcers on endoscopy, and have cardiopulmonary function tolerating the radiotherapy boost, a second phase of radiotherapy will be planned using a new CT simulation and radiotherapy design.
  First Phase of Radiotherapy: Total dose of 2500 cGy in 5 fractions (500 cGy per fraction). Second Phase of Radiotherapy: Total dose of 2500 cGy in 10 fractions (250 cGy per fraction) The interval between the two phases of radiotherapy will be 28 days.
  Interventions: Drug: Induction chemoimmunotherapy; Radiation: Hypofractionated Radiation Therapy; Drug: Concurrent Chemotherapy
- Conventional fractionated CCRT group (Active Comparator): Patients in this group will receive a total dose of 5000 cGy in 25 fractions, with 200 cGy per fraction.
  Interventions: Drug: Induction chemoimmunotherapy; Radiation: Conventional Fractionated Radiation Therapy; Drug: Concurrent Chemotherapy

INTERVENTIONS:
Drug: Induction chemoimmunotherapy — All patients will receive two cycles of induction therapy with albumin-bound paclitaxel and cisplatin combined with toripalimab.
Radiation: Hypofractionated Radiation Therapy — All patients will receive hypofractionated radiotherapy once daily, five days per week, followed by a boost. Three weeks after the completion of the first phase of hypofractionated radiotherapy, tumor response and cardiopulmonary function will be evaluated. For patients who achieve a partial response, have no deep esophageal ulcers on endoscopy, and have cardiopulmonary function tolerating the radiotherapy boost, a second phase of radiotherapy will be planned using a new CT simulation and radiotherapy design.
  First Phase of Radiotherapy: Total dose of 2500 cGy in 5 fractions (500 cGy per fraction) Second Phase of Radiotherapy: Total dose of 2500 cGy in 10 fractions (250 cGy per fraction) The interval between the two phases of radiotherapy will be 28 days.
  Arms: Hypofractionated CCRT group
Radiation: Conventional Fractionated Radiation Therapy — Patients will receive a total dose of 5000 cGy in 25 fractions, with 200 cGy per fraction.
  Arms: Conventional fractionated CCRT group
Drug: Concurrent Chemotherapy — Capecitabine oral administration, 1000 mg/m², twice daily

SUMMARY:
This is a prospective, open-label, randomized phase II clinical trial designed to compare the efficacy and toxicity of hypofractionated concurrent chemoradiotherapy versus conventional fractionated concurrent chemoradiotherapy following induction chemoimmunotherapy in patients with unresectable locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized phase II clinical trial designed to compare the efficacy and toxicity of hypofractionated concurrent chemoradiotherapy versus conventional fractionated concurrent chemoradiotherapy following induction chemoimmunotherapy in patients with unresectable locally advanced esophageal squamous cell carcinoma. In this study, patients will receive induction therapy with albumin-bound paclitaxel and cisplatin combined with toripalimab. After induction therapy, they will be randomly assigned to receive either definitive hypofractionated concurrent chemoradiotherapy or conventional fractionated concurrent chemoradiotherapy. Following the completion of treatment, patients will undergo regular follow-up to assess efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed diagnosis of esophageal squamous cell carcinoma;
* Evaluated as unresectable locally advanced esophageal squamous cell carcinoma by endoscopic ultrasound, imaging studies including esophagography, CT of the neck, chest, and upper abdomen, MRI of the neck and chest, whole-body bone scan, or PET/CT, with staging in the range of II-IVB (stage IVB limited to celiac lymph node or supraclavicular lymph node metastasis);
* Male or female aged 18 to 80 years;
* Eligible for oral drug therapy;
* No prior chemotherapy, radiotherapy, surgery, targeted therapy, or immunotherapy;
* Tumor sample requirement: Must provide adequate unstained, archived tumor tissue samples for analysis;
* Expected survival ≥12 weeks;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
* Postmenopausal women, or women with a negative urine or serum pregnancy test within 14 days before the study drug administration;
* Women must not be breastfeeding;
* Organ and bone marrow function must meet the following criteria: Forced expiratory volume in 1 second (FEV1) ≥1000 mL; Absolute neutrophil count ≥1.5 × 10^9/L; Platelets ≥100 × 10^9/L; Hemoglobin ≥90 g/L; Estimated glomerular filtration rate (eGFR) ≥50 mL/min based on the Cockcroft-Gault formula (Cockcroft and Gault, 1976); Serum bilirubin ≤1.5 × the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN;
* Signed and dated informed consent must be provided before participation in any study procedures.

Exclusion Criteria:

Exclusion Criteria for Induction Treatment:

* Participation in another clinical trial, unless it is an observational (non-interventional) study;
* Use of immunosuppressive drugs within 28 days prior to the first infusion of Toripalimab, excluding physiological doses of intranasal inhaled corticosteroids, prednisone ≤10 mg/day, or equivalent systemic corticosteroids;
* Prior use of any anti-PD-1 or anti-PD-L1 antibody;
* Major surgery within 4 weeks prior to entering the study (excluding vascular access procedures);
* A history of autoimmune disease within the past 2 years;
* Active or a history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis);
* History of primary immunodeficiency;
* History of organ transplantation requiring immunosuppressive treatment;
* Uncontrolled complications, including but not limited to persistent or active infections, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, arrhythmias, active peptic ulcer disease or gastritis, active bleeding disorders, including any known HBsAg-positive patients with HBV DNA >500 IU/ml, hepatitis C, or HIV, or any psychiatric or social conditions that would impair the ability to comply with study requirements or harm the patient's ability to provide written informed consent;
* Receipt of a live attenuated vaccine within 30 days prior to study initiation or within 30 days after receiving Toripalimab;
* History of another primary malignancy within 5 years prior to the initiation of Toripalimab treatment, excluding adequately treated skin basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix;
* Pregnancy, breastfeeding women, or men and women of reproductive potential who are not using effective contraception.

Exclusion Criteria for Concurrent Chemoradiotherapy After Induction Treatment:

* Development of distant metastasis (excluding celiac lymph node or supraclavicular lymph node metastasis);
* Development of local regional progression, with the radiation oncologist assessing that the patient cannot receive definitive chemoradiotherapy due to normal tissue dose limitations;
* PS score of 2-4;
* Any of the following organ and bone marrow dysfunction criteria: FEV1 <1000 mL; absolute neutrophil count <1.5 × 10^9/L; platelets <100 × 10^9/L; hemoglobin <90 g/L; serum creatinine clearance <50 mL/min according to the Cockcroft-Gault formula (Cockcroft & Gault, 1976); serum bilirubin >1.5 times the upper limit of normal (ULN); ALT and AST >2.5 times ULN.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2029-04-04 (Estimated); Study Completion 2029-04-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 2 years
  The proportion of patients who remain free from disease progression during a defined period after treatment initiation.

SECONDARY OUTCOMES:
Overall survival rate | 2 years
  The proportion of patients who are still alive after a specified period of time, regardless of disease progression or relapse.
Clinical response rate | 2 months after radiotherapy
  The percentage of patients who had partial remission or complete remission after therapy
Rate of grade 3 or higher toxicities | 1 year after therapy
  The percentage of patients who develop grade 3 or higher toxicities. The toxicities are evaluated based on Common Terminology Criteria for Adverse Events version 5.0. The values range from 1 to 5. A higher score means a worse outcome.
Distant metastasis-free survival rate | 2 years
Locoregional recurrence-free survival rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang X, Han W, Zhang W, Wang X, Ge X, Lin Y, Zhou H, Hu M, Wang W, Liu K, Lu J, Qie S, Zhang J, Deng W, Wang L, Han C, Li M, Zhang K, Li L, Wang Q, Shi H, Yu Z, Zhao Y, Sun X, Shi Y, Pang Q, Zhou Z, Liang J, Chen D, Feng Q, Bi N, Zhang T, Deng L, Wang W, Liu W, Wang J, Zhai Y, Wang J, Chen W, Chen J, Xiao Z; Jing-Jin-Ji Esophageal and Esophagogastric Cancer Radiotherapy Oncology Group (3JECROG). Effectiveness of S-1-Based Chemoradiotherapy in Patients 70 Years and Older With Esophageal Squamous Cell Carcinoma: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2312625. doi: 10.1001/jamanetworkopen.2023.12625. PMID 37195667
- [Background] Guo S, Liu F, Liu H, Wu Y, Zhang X, Ye W, Luo G, Li Q, Chen N, Hu N, Wang B, Zhang J, Lin M, Feng H, Qiu B. A Prospective Phase II Study of Simultaneous Modulated Accelerated Radiotherapy Concurrently With CDDP/S1 for Esophageal Squamous Cell Carcinoma in the Elderly. Front Oncol. 2021 Nov 25;11:760631. doi: 10.3389/fonc.2021.760631. eCollection 2021. PMID 34900709
- [Background] Song YP, Ma JB, Hu LK, Zhou W, Chen EC, Zhang W. Phase I/II study of hypofractioned radiation with three-dimensional conformal radiotherapy for clinical T3-4N0-1M0 stage esophageal carcinoma. Technol Cancer Res Treat. 2011 Feb;10(1):25-30. doi: 10.7785/tcrt.2012.500176. PMID 21214285
- [Background] Hulshof MCCM, Geijsen ED, Rozema T, Oppedijk V, Buijsen J, Neelis KJ, Nuyttens JJME, van der Sangen MJC, Jeene PM, Reinders JG, van Berge Henegouwen MI, Thano A, van Hooft JE, van Laarhoven HWM, van der Gaast A. Randomized Study on Dose Escalation in Definitive Chemoradiation for Patients With Locally Advanced Esophageal Cancer (ARTDECO Study). J Clin Oncol. 2021 Sep 1;39(25):2816-2824. doi: 10.1200/JCO.20.03697. Epub 2021 Jun 8. PMID 34101496
- [Background] Minsky BD, Neuberg D, Kelsen DP, Pisansky TM, Ginsberg RJ, Pajak T, Salter M, Benson AB 3rd. Final report of Intergroup Trial 0122 (ECOG PE-289, RTOG 90-12): Phase II trial of neoadjuvant chemotherapy plus concurrent chemotherapy and high-dose radiation for squamous cell carcinoma of the esophagus. Int J Radiat Oncol Biol Phys. 1999 Feb 1;43(3):517-23. doi: 10.1016/s0360-3016(98)00463-5. PMID 10078631
- [Background] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Background] Kojima T, Shah MA, Muro K, Francois E, Adenis A, Hsu CH, Doi T, Moriwaki T, Kim SB, Lee SH, Bennouna J, Kato K, Shen L, Enzinger P, Qin SK, Ferreira P, Chen J, Girotto G, de la Fouchardiere C, Senellart H, Al-Rajabi R, Lordick F, Wang R, Suryawanshi S, Bhagia P, Kang SP, Metges JP; KEYNOTE-181 Investigators. Randomized Phase III KEYNOTE-181 Study of Pembrolizumab Versus Chemotherapy in Advanced Esophageal Cancer. J Clin Oncol. 2020 Dec 10;38(35):4138-4148. doi: 10.1200/JCO.20.01888. Epub 2020 Oct 7. PMID 33026938
- [Background] Gaspar LE, Winter K, Kocha WI, Coia LR, Herskovic A, Graham M. A phase I/II study of external beam radiation, brachytherapy, and concurrent chemotherapy for patients with localized carcinoma of the esophagus (Radiation Therapy Oncology Group Study 9207): final report. Cancer. 2000 Mar 1;88(5):988-95. PMID 10699886
- [Background] Chen Y, Ye J, Zhu Z, Zhao W, Zhou J, Wu C, Tang H, Fan M, Li L, Lin Q, Xia Y, Li Y, Li J, Jia H, Lu S, Zhang Z, Zhao K. Comparing Paclitaxel Plus Fluorouracil Versus Cisplatin Plus Fluorouracil in Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Cancer: A Randomized, Multicenter, Phase III Clinical Trial. J Clin Oncol. 2019 Jul 10;37(20):1695-1703. doi: 10.1200/JCO.18.02122. Epub 2019 Mar 28. PMID 30920880
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338